CLINICAL TRIAL: NCT06953531
Title: The Effect of Three Different Methods Used During Blood Collection in Children on Pain, Fear and Procedure Time
Brief Title: The Effect of Methods Used During Blood Collection on Pain and Fear in Children
Acronym: pain and fear
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice ŞEN (Other)
Responsible Party: Sponsor-Investigator, Hatice ŞEN, Research Assistant, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: University Mersin
Record Dates: First submitted 2025-04-20; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pain; Fear
Keywords: Blood collection process in children; Nursing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Local Skin Cooling Device Group (Experimental): Participants are given a cold application using a local skin cooling device just before the blood collection process.
  Interventions: Device: Cold Application (Local Skin Cooling Device)
- Bubble Machine Group (Experimental): During the blood collection process, participants are entertained with the bubble machine.
  Interventions: Behavioral: Distraction Method (Bubble Machine)
- Simulative Toy Group (Experimental): During the blood collection process, participants are distracted with a simulative toy.
  Interventions: Behavioral: Distraction Method (Simulative Toy)
- Control Group (No Intervention): Participants are not subjected to any intervention during the blood collection process.

INTERVENTIONS:
Device: Cold Application (Local Skin Cooling Device) — Immediately before the blood collection procedure, cold application will be made to the area with a local skin cooling device.
  Arms: Local Skin Cooling Device Group
Behavioral: Distraction Method (Bubble Machine) — A bubble machine will be used to distract children during the blood collection process.
  Arms: Bubble Machine Group
Behavioral: Distraction Method (Simulative Toy) — A simulative toy will be used to distract children during the blood collection process.
  Arms: Simulative Toy Group

SUMMARY:
The effect of three different methods (local skin cooling device, bubble machine, simulative toy) that will be used during the blood collection procedure on pain, fear and procedure time will be investigated in pain-sensitive 6-12 age group children.

DETAILED DESCRIPTION:
Children are usually admitted to the hospital for diagnosis, treatment or follow-up at an early stage of their lives and are subjected to various invasive procedures during this process. Blood collection is one of the interventions that are repeated many times by children during diagnosis and treatment, causing a feeling of pain and fear. Although bloodletting may seem like a minor procedure, it is considered a source of great fear by children and therefore turns into an unpleasant experience by both children and their families.

Pain management is both an ethical obligation and a child's right, which should be done by focusing on the needs and preferences of children and their parents, requires accurate and effective planning. Nonpharmacological treatment methods used in pain management in children are classified into three groups: physical, supportive and cognitive-behavioral methods. The use of Coolsense, a local skin cooling device, is a method that can be used in this sense in terms of its rapid effect. Coolsense; it is a hand-held device that has an effect in as little as five seconds, does not contain chemicals, has a temperature-controlled head, can be stored in the freezer of refrigerators and used repeatedly. Among the advantages of the device are that it is easy to use, it is applied to a small area and it is easy to Decipher whether it is at the right temperature from the light burning on it. The most preferred method among cognitive-behavioral methods is the method of diverting attention Decently. The method of diverting attention is divided into two as active and passive methods. One of the methods of attracting active attention is the use of toys. One of these toys is a bubble machine. The bubble machine is a toy with the ability to produce a large number of bubbles at the same time with its multi-hole design. With this toy, the child focuses on the bubbles that come out through the bubble machine, and not on the painful process, so his attention is diverted from the blood collection process. Another one of the toys is a simulative toy. Simulative toy; it is a toy that can show realistic and vivid features, contains sensors sensitive to touch and movement, breathes, can open and close its eyes, can move its head and body, and at the same time make sounds as if it were real. With these features, it can be effective in reducing pain and fear by ensuring that children's attention is diverted from the painful procedure. It is thought that three different methods (local skin cooling device, bubble machine, simulative toy) that will be used during the blood collection procedure in pain-sensitive 6-12 age group children may have a positive effect on pain, fear and procedure time.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between the ages of 6 and 12.
* The child's WB-YİDÖ score must be 0 before the blood collection procedure.
* The child must be willing to participate in the study and sign the Informed Consent Form/Written Consent Form.
* The child must be able to speak Turkish.
* The child must not have a mental disability and must be able to use their arms functionally.
* The child must not have used sedatives, analgesics, or narcotics within 6 hours prior to admission to the blood collection unit.
* The child's body temperature must be below 38 °C at the time of admission to the blood collection unit.
* The child must have undergone blood collection procedures before.
* The child must not be afraid of the simulation toy.

Exclusion Criteria:

* Failure to sign the Informed Consent Form/Written Consent Form.
* The child has a disease that causes chronic pain.
* The child has vision or hearing problems.
* Deterioration of skin integrity in the blood collection area or in the area where the local skin cooling device will be applied.
* Presence of nerve damage in the area where blood will be drawn.
* Having sensory motor deficit, diabetes, peripheral vascular disease (e.g., Raynaud's syndrome), neuropathy, or sickle cell anemia.
* The child has an allergy to the simulative toy.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Facial Expressions Rating Scale | At the time of blood collection (0 minutes) and 5 minutes after the procedure
  The Wong-Baker Facial Expressions Rating Scale will be used to assess the pain levels of children during the blood collection procedure and 5 minutes after the procedure. The scale includes six facial expressions representing increasing levels of pain, scored from 0 (no pain) to 5 or 10 (severe pain), depending on the version used.
Children's Fear Scale | Immediately before and during the blood collection procedure.
  The Child Fear Scale, which is suitable for children aged 3 to 16, will be used to assess the level of fear and anxiety experienced by the child before and during the blood collection. The scale consists of five facial expressions scored from 0 (no fear and anxiety) to 4 (highest fear and anxiety), and can be administered by children, parents, or researchers.

IPD SHARING:
Plan to Share IPD: No